CLINICAL TRIAL: NCT03723278
Title: Single-centre, Single-blind, Randomized, Controlled, Cross-over Study to Analyze the Influence of Nitric Oxide on Flow Mediated Dilation
Brief Title: Influence of Nitric Oxide on Flow Mediated Dilation
Status: Completed | Type: Observational
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Principal Investigator, Roland E. Schmieder, Principal Investigator, University of Erlangen-Nürnberg Medical School
Other Study IDs: CRC2018UNEX
Record Dates: First submitted 2018-10-11; First posted 2018-10-29 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: FMD - Flow Mediated Dilation
Keywords: nitric oxide

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy individuals: Young, male and healthy volunteers without any significant disease

SUMMARY:
Flow-mediated vasodilation (FMD) has become one of the most widely assessed parameter to analyze endothelial function. The peripheral endothelial function as assessed by FMD correlates with coronary artery endothelial function and moreover, impaired FMD has been revealed to be good predictor for cardiovascular events in patients beyond cardiovascular risk factors and in patients with coronary artery disease.

This non-invasive technique measures the ability of the arteries to respond with endothelial release of vasoactive factors during reactive hyperemia. In this study the goal is to analyze in a clinical trial to what extend nitric oxide contribute to FMD by measuring FMD before and after blocking the release of nitric oxide. FMD is measured using a semi-automatic device named UNEX, recently developed in Japan. This semi-automatic ultrasound system represents a new development that overcomes the limitation of classic systems.

The hypothesis of this study is that FMD response is mostly nitric oxide dependent. To prove this hypothesis, overall 20 healthy male volunteers are included in this study. Total duration of this study for each volunteer is 2-4 weeks with total 3 visits at the Clinical Research Unit (CRC) of the Department of Nephrology, University of Erlangen-Nuremberg.

This study is important to better understand the mechanism of any kind of impaired FMD by cardiovascular risk factors and diseases and to better interpret impaired FMD assessed by UNEX.

DETAILED DESCRIPTION:
The assessment of endothelial function is crucial, as its dysfunction is described as a key pathological condition associated with many diseases leading to arteriosclerosis. Flow-mediated vasodilation (FMD) has become one of the most widely assessed parameter to analyze endothelial function. Celermajer et al. was the first to measure the FMD-response in vivo by ultrasound. This non-invasive technique measures the ability of the arteries to respond with endothelial release of vasoactive factors during reactive hyperemia.

The peripheral endothelial function as assessed by FMD correlates with coronary artery endothelial function. Impaired FMD has been revealed to be good predictor for cardiovascular events in patients beyond cardiovascular risk factors and in patients with coronary artery disease. It is also predictive for the extent and severity of coronary atherosclerosis.

Beyond the predictive nature of FMD, several studies have been reported on the effect of pharmacologic or physiologic interventions on FMD. For example weight loss and exercise increased FMD in overweight and obese patients with coronary heart disease.

Impaired FMD is mainly characterized by reduced bioavailability of different vasodilators due to oxidative stress. Of these vasodilators nitric oxide plays the major role, but its contribution to FMD is inconclusive. Studies to clarify the role of nitric oxide on FMD have been done with various methods, which require extensive training and standardization. Operator, study preparation, image acquisition and site selection, sphygmomanometer probe position, cuff occlusion time, the accurate use of edge-detection software as well as the correct characterization of the FMD response are all factors, which influence FMD measurement.

In this study the goal is to analyze in a clinical trial to what extent nitric oxide contribute to FMD by measuring FMD before and after blocking the release of nitric oxide. FMD is measured using a semi-automatic device named UNEX, recently developed in Japan. FMD measurements using UNEX implement the standards described in guidelines. This semi-automatic ultrasound system using an H-type ultrasound probe represents a new development that overcomes the limitation of classic systems (in particular the investigator-dependency of conventional, "hand-held" FMD measurements). This system comprised a 7.5-megahertz linear array transducer and a novel stereotactic probe-holding device (UNEX Co., Nagoya, Japan). Another advantage of this device is the continuous recording of B-mode images and A-mode waves of the artery in the longitudinal plane, so that continuous measurement of arterial diameter in the 4.5 min following cuff deflation occurs. A meta-analysis described that the nitric oxide dependency of the FMD response was the most in studies with FMD measurements at brachial artery with distal placement of the cuff and 5-minute occlusion. These criteria are fulfilled by UNEX. However, no data on nitric oxide dependency are available in the literature. Finally, this semi-automatic assessment of FMD has been shown to improve the precision and repeatability of the measurements.

The hypothesis of this study is that FMD response is mostly nitric oxide dependent and this could not be proven so far due to less sensitive conventional tool of FMD measurement.

ELIGIBILITY:
Inclusion Criteria:

* Young, male and healthy volunteers without any significant disease
* Age of 18 and 45 years old
* Informed consent has to be given in written form

Exclusion Criteria:

* Uncontrolled hypertension or blood pressure >160/100 mmHg
* Known Diabetes mellitus or fasting plasma glucose >126mg/dl
* Subjects having any chronic treatment
* Drug or alcohol abuse
* Allergies or intolerance against the substances used in the study
* Smokers or subjects had stopped smoking <1 year
* Participation in another clinical study within 30 days prior to V1
* Subject who do not give written consent, that pseudonymous data will be transferred in line with the duty of documentation and the duty of notification according to § 12 and § 13 Good Clinical Practice-V

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: * Young, male and healthy volunteers without any significant disease
  * Age of 18 and 45 years old
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2018-11-14 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Percent change of flow mediated dilation | 1 week after study inclusion
  Percent change of flow mediated dilation (UNEX EF) in Response to L-NMMA/Saline infusion
Percent change of flow mediated dilation | 2 weeks after study inclusion
  Percent change of flow mediated dilation (UNEX EF) in Response to L-NMMA/Saline infusion

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Research Center, Department of Nephrology and Hypertension, University of Erlangen-Nuremberg, Erlangen, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Makimattila S, Virkamaki A, Groop PH, Cockcroft J, Utriainen T, Fagerudd J, Yki-Jarvinen H. Chronic hyperglycemia impairs endothelial function and insulin sensitivity via different mechanisms in insulin-dependent diabetes mellitus. Circulation. 1996 Sep 15;94(6):1276-82. doi: 10.1161/01.cir.94.6.1276. PMID 8822980
- [Background] Panza JA, Quyyumi AA, Brush JE Jr, Epstein SE. Abnormal endothelium-dependent vascular relaxation in patients with essential hypertension. N Engl J Med. 1990 Jul 5;323(1):22-7. doi: 10.1056/NEJM199007053230105. PMID 2355955
- [Background] Celermajer DS, Sorensen KE, Gooch VM, Spiegelhalter DJ, Miller OI, Sullivan ID, Lloyd JK, Deanfield JE. Non-invasive detection of endothelial dysfunction in children and adults at risk of atherosclerosis. Lancet. 1992 Nov 7;340(8828):1111-5. doi: 10.1016/0140-6736(92)93147-f. PMID 1359209
- [Background] Anderson TJ, Uehata A, Gerhard MD, Meredith IT, Knab S, Delagrange D, Lieberman EH, Ganz P, Creager MA, Yeung AC, et al. Close relation of endothelial function in the human coronary and peripheral circulations. J Am Coll Cardiol. 1995 Nov 1;26(5):1235-41. doi: 10.1016/0735-1097(95)00327-4. PMID 7594037
- [Background] Yeboah J, Crouse JR, Hsu FC, Burke GL, Herrington DM. Brachial flow-mediated dilation predicts incident cardiovascular events in older adults: the Cardiovascular Health Study. Circulation. 2007 May 8;115(18):2390-7. doi: 10.1161/CIRCULATIONAHA.106.678276. Epub 2007 Apr 23. PMID 17452608
- [Background] Neunteufl T, Katzenschlager R, Hassan A, Klaar U, Schwarzacher S, Glogar D, Bauer P, Weidinger F. Systemic endothelial dysfunction is related to the extent and severity of coronary artery disease. Atherosclerosis. 1997 Feb 28;129(1):111-8. doi: 10.1016/s0021-9150(96)06018-2. PMID 9069525
- [Background] Ades PA, Savage PD, Lischke S, Toth MJ, Harvey-Berino J, Bunn JY, Ludlow M, Schneider DJ. The effect of weight loss and exercise training on flow-mediated dilatation in coronary heart disease: a randomized trial. Chest. 2011 Dec;140(6):1420-1427. doi: 10.1378/chest.10-3289. Epub 2011 Jul 21. PMID 21778256
- [Background] Joannides R, Haefeli WE, Linder L, Richard V, Bakkali EH, Thuillez C, Luscher TF. Nitric oxide is responsible for flow-dependent dilatation of human peripheral conduit arteries in vivo. Circulation. 1995 Mar 1;91(5):1314-9. doi: 10.1161/01.cir.91.5.1314. PMID 7867167
- [Background] Green DJ, Dawson EA, Groenewoud HM, Jones H, Thijssen DH. Is flow-mediated dilation nitric oxide mediated?: A meta-analysis. Hypertension. 2014 Feb;63(2):376-82. doi: 10.1161/HYPERTENSIONAHA.113.02044. Epub 2013 Nov 25. PMID 24277765
- [Background] Iguchi T, Takemoto Y, Shimada K, Matsumoto K, Nakanishi K, Otsuka K, Hyodo E, Hirohashi K, Tahara A, Yoshiyama M. Simultaneous assessment of endothelial function and morphology in the brachial artery using a new semiautomatic ultrasound system. Hypertens Res. 2013 Aug;36(8):691-7. doi: 10.1038/hr.2013.35. Epub 2013 Apr 18. PMID 23595043
- [Background] Tomiyama H, Kohro T, Higashi Y, Takase B, Suzuki T, Ishizu T, Ueda S, Yamazaki T, Furumoto T, Kario K, Inoue T, Koba S, Watanabe K, Takemoto Y, Hano T, Sata M, Ishibashi Y, Node K, Maemura K, Ohya Y, Furukawa T, Ito H, Ikeda H, Yamashina A. Reliability of measurement of endothelial function across multiple institutions and establishment of reference values in Japanese. Atherosclerosis. 2015 Oct;242(2):433-42. doi: 10.1016/j.atherosclerosis.2015.08.001. Epub 2015 Aug 5. PMID 26291496